CLINICAL TRIAL: NCT02761447
Title: Effectivity of Differences Therapies on Central Nerve System for Pain, Phantom, Disability and Quality of Life in Amputees
Brief Title: Effectivity of Motor Imagery and MirrorTherapy in Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD,, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI15_25
Record Dates: First submitted 2016-04-21; First posted 2016-05-04 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Amputees
Keywords: Motor control Laterality; Pain Perception; Lower Extremity; Complementary Therapies; Physical Therapy Modalities
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Traditional and Motor Imaginary Program (Experimental): Amputees patients also conservative protocol will undergo physiotherapy techniques work Motor Imaginary Program, based on a system of two videos that allow the patient to recreate the "normal" way. The first video will include two sequences of a harmonic gear that will allow the patient to examine, with the physiotherapist, the characteristics of the different body segments involved in locomotion and place the member in space. The second video include an analysis in five phases. This protocol will be applied 3 days a week (25-30minutos) for one month.
  Interventions: Other: Treatment Traditional and Imaginary Motor Program
- Treatment Traditional and Mirror Therapy (Active Comparator): Amputees patients also conservative protocol will undergo physical therapy techniques mirror therapy work. The protocol will consist of mirror therapy sessions three days a week (25-30 minutes) for a month, where participants will move the intact limb looking in the mirror and imagining the movement of the limb with phantom sensation.
  Interventions: Other: Treatment Traditional and Mirror Therapy

INTERVENTIONS:
Other: Treatment Traditional and Imaginary Motor Program — Amputees patients also conservative protocol will undergo physiotherapy techniques work Imaginary Motor. The first video will include two sequences of a harmonic gear that will allow the patient to examine, with the physiotherapist, the characteristics of the different body segments involved in locomotion and place the member in space. The second video include an analysis in five phases: a) relaxation of Benson, b) phase external imagination where cycles of normal running on a video provided by the physiotherapist, c) phase internal imagination where the patient will identify the problem discussed compared with the normal course presented in the video, d) recreation of images in the first person made an e normalized locomotion) closing his eyes, prompted the patient to mentally recreate sequences normal gait and analyzed and subsequently verbalize differences of these with respect to their own way of getting around.
  Arms: Treatment Traditional and Motor Imaginary Program
Other: Treatment Traditional and Mirror Therapy — Amputees patients also conservative protocol will undergo physiotherapy techniques mirror therapy work. The protocol will consist of mirror therapy sessions three days a week (25-30 minutes) for a month, where participants will move the intact limb looking in the mirror and imagining the movement of the limb with phantom sensation.
  Arms: Treatment Traditional and Mirror Therapy

SUMMARY:
This study evaluates the effectiveness of imagery motor on phantom pain and amputation process

DETAILED DESCRIPTION:
The expected increase in the number of amputations in the coming decades requires special attention to the common effect after called phantom limb amputation. That term refers to the phenomena covering the sensations that occur in the affected limb and whose prevalence rate is an important part of amputees subjects. Developed theories about their origin focus their attention on the central nervous system and the peripheral nervous system. Thus, the imaginary movement is a complex cognitive, sensory and proprioceptive process leading to a mental representation of movement and it is a widely used technique in neurological rehabilitation and complex pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the stump area ≥ 3 months, no intermittent
2. Have three months elapsed amputation,
3. Submit subjective sensation of phantom limb not blinking

Exclusion Criteria:

* Clinical signs of radiculopathy.
* Lumbar stenosis, fibromyalgia, spondylolisthesis.
* History of spinal surgery.
* Corticosteroid therapy in the past two weeks.
* Disease of the central nervous system or peripheral.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Changes from Baseline Numerical Rating Scale at one month. Changes from Baseline Numerical Rating Scale at three months

SECONDARY OUTCOMES:
McGiII Pain Questionnaire (MPQ) | Changes from Baseline McGiII Pain Questionnaire at one month. Changes from Baseline McGiII Pain Questionnaire at three months
The Vividness of Visual Imagery Questionnaire | Changes from Baseline Vividness of Visual Imagery Questionnaire at one month and three months
Beck Depression Inventory | Changes from Baseline Beck Depression Inventory at one month. Changes from Baseline Beck Depression Inventory at three months
Neuropathic Pain Questionnaire (DN4) | Changes from Baseline Neuropathic Pain Questionnaire at one month. Changes from Baseline Neuropathic Pain Questionnaire at three months
Pressure Algometer (kg/cm2) | Changes from Baseline Pressure Algometer at one month. Changes from Baseline Pressure Algometer at three months
  Pressure algometer in lumbar pain, amputated limb and health limb
West-Haven-Yale Multidimensional Pain Inventory | Changes from Baseline West-Haven-Yale Multidimensional Pain Inventory at one month. Changes from Baseline West-Haven-Yale Multidimensional Pain Inventory at three months
The Barthel Index of ADLs | Changes from Baseline Barthel Index of ADLs at one month. Changes from Baseline Barthel Index of ADLs at three months
Instrumental Activities of Daily Living Scale (IADL) | Changes from Baseline Instrumental Activities of Daily Living Scale at one month. Changes from Baseline Instrumental Activities of Daily Living Scale at three months
The Functional Independence Measure Scale (FIM) | Changes from Baseline Functional Independence Measure Scale at one month. Changes from Baseline Functional Independence Measure Scale at three months
Quality of Life Questionnaire scoring (SF36) | Changes from Baseline Quality of Life Questionnaire Scoring at one month. Changes from Baseline Quality of Life Questionnaire Scoring at three months
Multidimensional Body Self Relations Questionnaire (MBSRQ) | Changes from Baseline Multidimensional Body Self Relations Questionnaire at one month. Changes from Baseline Multidimensional Body Self Relations Questionnaire at three months
Tampa Scale for Kinesiophobia (TSK) | Changes from Baseline Tampa Scale for Kinesiophobia at one month. Changes from Baseline Tampa Scale for Kinesiophobia at three months
Pain Catastrophizing Scale (PCS) | Changes from Baseline Pain Catastrophizing Scale at one month. Changes from Baseline Pain Catastrophizing Scale at three months
Pain Management Inventory | Changes from Baseline Pain Management Inventory at one month. Changes from Baseline Pain Management Inventory at three months

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Hospital de Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Ephraim PL, Wegener ST, MacKenzie EJ, Dillingham TR, Pezzin LE. Phantom pain, residual limb pain, and back pain in amputees: results of a national survey. Arch Phys Med Rehabil. 2005 Oct;86(10):1910-9. doi: 10.1016/j.apmr.2005.03.031. PMID 16213230
- [Background] Raichle KA, Hanley MA, Molton I, Kadel NJ, Campbell K, Phelps E, Ehde D, Smith DG. Prosthesis use in persons with lower- and upper-limb amputation. J Rehabil Res Dev. 2008;45(7):961-72. doi: 10.1682/jrrd.2007.09.0151. PMID 19165686
- [Background] Foell J, Bekrater-Bodmann R, Flor H, Cole J. Phantom limb pain after lower limb trauma: origins and treatments. Int J Low Extrem Wounds. 2011 Dec;10(4):224-35. doi: 10.1177/1534734611428730. PMID 22184752
- [Background] Seidel S, Kasprian G, Furtner J, Schopf V, Essmeister M, Sycha T, Auff E, Prayer D. Mirror therapy in lower limb amputees--a look beyond primary motor cortex reorganization. Rofo. 2011 Nov;183(11):1051-7. doi: 10.1055/s-0031-1281768. Epub 2011 Sep 28. PMID 21959885
- [Background] Flor H. Maladaptive plasticity, memory for pain and phantom limb pain: review and suggestions for new therapies. Expert Rev Neurother. 2008 May;8(5):809-18. doi: 10.1586/14737175.8.5.809. PMID 18457537
- [Background] Bosmans JC, Geertzen JH, Post WJ, van der Schans CP, Dijkstra PU. Factors associated with phantom limb pain: a 31/2-year prospective study. Clin Rehabil. 2010 May;24(5):444-53. doi: 10.1177/0269215509360645. PMID 20442256
- [Background] Priganc VW, Stralka SW. Graded motor imagery. J Hand Ther. 2011 Apr-Jun;24(2):164-8; quiz 169. doi: 10.1016/j.jht.2010.11.002. Epub 2011 Feb 9. PMID 21306870
- [Background] Janig W, Baron R. Complex regional pain syndrome: mystery explained? Lancet Neurol. 2003 Nov;2(11):687-97. doi: 10.1016/s1474-4422(03)00557-x. PMID 14572737
- [Background] McCabe CS, Haigh RC, Ring EF, Halligan PW, Wall PD, Blake DR. A controlled pilot study of the utility of mirror visual feedback in the treatment of complex regional pain syndrome (type 1). Rheumatology (Oxford). 2003 Jan;42(1):97-101. doi: 10.1093/rheumatology/keg041. PMID 12509620
- [Background] Pleger B, Tegenthoff M, Ragert P, Forster AF, Dinse HR, Schwenkreis P, Nicolas V, Maier C. Sensorimotor retuning [corrected] in complex regional pain syndrome parallels pain reduction. Ann Neurol. 2005 Mar;57(3):425-9. doi: 10.1002/ana.20394. PMID 15732114
- [Background] Maihofner C, Handwerker HO, Neundorfer B, Birklein F. Patterns of cortical reorganization in complex regional pain syndrome. Neurology. 2003 Dec 23;61(12):1707-15. doi: 10.1212/01.wnl.0000098939.02752.8e. PMID 14694034
- [Background] Mercier C, Sirigu A. Training with virtual visual feedback to alleviate phantom limb pain. Neurorehabil Neural Repair. 2009 Jul-Aug;23(6):587-94. doi: 10.1177/1545968308328717. Epub 2009 Jan 26. PMID 19171946
- [Background] Dickstein R, Deutsch JE. Motor imagery in physical therapist practice. Phys Ther. 2007 Jul;87(7):942-53. doi: 10.2522/ptj.20060331. Epub 2007 May 1. PMID 17472948
- [Background] Berthelot JM. Current management of reflex sympathetic dystrophy syndrome (complex regional pain syndrome type I). Joint Bone Spine. 2006 Oct;73(5):495-9. doi: 10.1016/j.jbspin.2005.11.022. Epub 2006 Jun 30. PMID 16837228
- [Background] Daly AE, Bialocerkowski AE. Does evidence support physiotherapy management of adult Complex Regional Pain Syndrome Type One? A systematic review. Eur J Pain. 2009 Apr;13(4):339-53. doi: 10.1016/j.ejpain.2008.05.003. Epub 2008 Jul 10. PMID 18619873
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Lotze M, Grodd W, Birbaumer N, Erb M, Huse E, Flor H. Does use of a myoelectric prosthesis prevent cortical reorganization and phantom limb pain? Nat Neurosci. 1999 Jun;2(6):501-2. doi: 10.1038/9145. No abstract available. PMID 10448212
- [Background] Flor H, Denke C, Schaefer M, Grusser S. Effect of sensory discrimination training on cortical reorganisation and phantom limb pain. Lancet. 2001 Jun 2;357(9270):1763-4. doi: 10.1016/S0140-6736(00)04890-X. PMID 11403816
- [Background] Hovington CL, Brouwer B. Guided motor imagery in healthy adults and stroke: does strategy matter? Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):851-7. doi: 10.1177/1545968310374190. Epub 2010 Sep 12. PMID 20834045
- [Background] Hwang S, Jeon HS, Yi CH, Kwon OY, Cho SH, You SH. Locomotor imagery training improves gait performance in people with chronic hemiparetic stroke: a controlled clinical trial. Clin Rehabil. 2010 Jun;24(6):514-22. doi: 10.1177/0269215509360640. Epub 2010 Apr 14. PMID 20392784
- [Background] Beaumont G, Mercier C, Michon PE, Malouin F, Jackson PL. Decreasing phantom limb pain through observation of action and imagery: a case series. Pain Med. 2011 Feb;12(2):289-99. doi: 10.1111/j.1526-4637.2010.01048.x. Epub 2011 Jan 28. PMID 21276185
- [Background] MacIver K, Lloyd DM, Kelly S, Roberts N, Nurmikko T. Phantom limb pain, cortical reorganization and the therapeutic effect of mental imagery. Brain. 2008 Aug;131(Pt 8):2181-91. doi: 10.1093/brain/awn124. Epub 2008 Jun 20. PMID 18567624
- [Background] Brodie EE, Whyte A, Niven CA. Analgesia through the looking-glass? A randomized controlled trial investigating the effect of viewing a 'virtual' limb upon phantom limb pain, sensation and movement. Eur J Pain. 2007 May;11(4):428-36. doi: 10.1016/j.ejpain.2006.06.002. Epub 2006 Jul 20. PMID 16857400
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Casale R, Alaa L, Mallick M, Ring H. Phantom limb related phenomena and their rehabilitation after lower limb amputation. Eur J Phys Rehabil Med. 2009 Dec;45(4):559-66. Epub 2009 Feb 26. PMID 20032915
- [Background] Sumitani M, Miyauchi S, McCabe CS, Shibata M, Maeda L, Saitoh Y, Tashiro T, Mashimo T. Mirror visual feedback alleviates deafferentation pain, depending on qualitative aspects of the pain: a preliminary report. Rheumatology (Oxford). 2008 Jul;47(7):1038-43. doi: 10.1093/rheumatology/ken170. Epub 2008 May 7. PMID 18463143
- [Background] Diers M, Christmann C, Koeppe C, Ruf M, Flor H. Mirrored, imagined and executed movements differentially activate sensorimotor cortex in amputees with and without phantom limb pain. Pain. 2010 May;149(2):296-304. doi: 10.1016/j.pain.2010.02.020. Epub 2010 Mar 31. PMID 20359825
- [Background] Brodie EE, Whyte A, Waller B. Increased motor control of a phantom leg in humans results from the visual feedback of a virtual leg. Neurosci Lett. 2003 May 1;341(2):167-9. doi: 10.1016/s0304-3940(03)00160-5. PMID 12686392
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273